CLINICAL TRIAL: NCT03397511
Title: Incorporating Financial Incentives to Increase Smoking Cessation Among Asian Americans Residing in New York City: A Feasibility Study
Brief Title: Incorporating Financial Incentives to Increase Smoking Cessation Among Asian Americans Residing in New York City
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00760
Record Dates: First submitted 2018-01-05; First posted 2018-01-12 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Smoking Cessation; Smoking, Cigarette
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual Care+Financial Incentive (Experimental): Smoking cessation counseling couples with financial incentives
  Interventions: Behavioral: Financial Incentives

INTERVENTIONS:
Behavioral: Financial Incentives — Baseline Interview, 2 Counseling Sessions at baseline and 2 weeks post baseline, and one follow up survey at one month

SUMMARY:
Financial incentives for motivating health change have been increasingly employed in various healthcare sectors. They can be a potentially effective approach to promote smoking behavioral change and increase the use of evidence-based counseling and pharmacotherapy. Smoking cessation randomized clinical trials (RCT) incorporating financial incentives have been conducted in different populations; however, there has not been a randomized clinical trial coupled with a financial incentive with Asian American cigarette smokers. The purpose of this pilot study is to examine the feasibility of implementing an incentivized smoking cessation program among Asian American smokers in New York City.

ELIGIBILITY:
Inclusion Criteria:

* Asian American
* current smoker who smokes at least 10 cigarettes daily (verified by a CO level of 8 ppm or above)
* New York City resident
* able to complete three month follow-up assessments in person, can provide a telephone number
* declining the use of Chantix for smoking cessation.

Exclusion Criteria:

* <18 years old
* pregnant
* cannot provide a telephone number, non-smokers or smokers that smoke fewer than 10 cigarettes daily, users of e-cigarettes or other tobacco products who are not interested in quitting smoking, marijuana users
* not a New York City resident
* unable to complete three month follow-up assessment in person
* unable to provide written consent
* agree to use Chantix for smoking cessation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Number of patients recruited by implementing Financial Incentive Smoking Cessation Program among Asian American Smokers | One Month
  Number of patients who complete incentive program

CONTACTS AND LOCATIONS:
Overall Officials: Donna Shelley, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided